CLINICAL TRIAL: NCT02786290
Title: The Zenflow Spring System Feasibility and Safety Study (ZEST)
Brief Title: The Zenflow Spring System Feasibility and Safety Study
Acronym: ZEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zenflow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0002
Record Dates: First submitted 2016-05-09; First posted 2016-05-30 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Receives intervention with the Zenflow Spring System.
  Interventions: Device: Zenflow Spring System

INTERVENTIONS:
Device: Zenflow Spring System — The Zenflow Spring is a nitinol urethral implant for the treatment of Lower Urinary Tract Symptoms (LUTS) that arise due to bladder outlet obstruction (BOO), secondary to the presence of Benign Prostatic Hypertrophy (BPH). The device is intended to be a permanent implant however it may be removed if necessary.

SUMMARY:
This is a First in Human study to assess the feasibility, safety and effectiveness of the Zenflow Spring System in relieving the symptoms of obstructive Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
The purpose of the Zenflow Study is to evaluate the feasibility and safety of a novel prostatic urethral implant for the treatment of Lower Urinary Tract Symptoms (LUTS) that arise due to bladder outlet obstruction (BOO), secondary to the presence of Benign Prostatic Hypertrophy (BPH). Effectiveness will also be measured. It is intended that the features of the Zenflow Spring will provide an effective office-based treatment and management therapy for BPH with little or no side effects.

ELIGIBILITY:
Inclusion Criteria:

1. 50 to 80 years of age
2. Baseline IPSS score > 13, and a baseline Quality of Life (Qol) question score > 3
3. Prostate volume 25 - 80 cc by Trans Rectal Ultrasound (TRUS), measured within past 90 days
4. Anterior prostatic urethral length 2.5 - 4.0 cm by cystoscopy, as measured from bladder neck to verumontanum. TRUS will be accepted as a primary screening measure.
5. Failed or intolerant to medication regimen for the treatment of LUTS.

Exclusion Criteria:

New Zealand only: A maximum of 5 participants in acute or chronic urinary retention may be included in the study provided they meet other entry criteria. Exclusion exemptions for these patients are described in 4a, 5a and they are exempt from #6.

Participants will be excluded from participating in this trial if they meet any of the following criteria:

1. Obstructive median prostatic lobe or high bladder neck
2. Urethral stricture, meatal stenosis, or bladder neck obstruction - either current, or recurrent requiring 2 or more dilatations
3. Elevated Prostate Specific Antigen (PSA) (age 50-70 PSA ≥4; age 70+ PSA ≥6.5) unless negative biopsy within last 3 months, or a positive biopsy
4. Post-void residual volume (PVR) > 250 ml, if not in acute retention 4a. No maximum post void residual volume required if patient in acute or chronic urinary retention. (New Zealand Only, up to 5 patients)
5. Peak urinary flow rate > 12 ml/second, with ≥ 125 ml voided volume at baseline. 5a. No maximum urinary flow or minimum voided volume required if participant in acute or chronic urinary retention. (New Zealand Only, up to 5 patients)
6. History of chronic urinary retention. (New Zealand Only, up to 5 patients)
7. History of neurogenic bladder
8. Compromised renal function (e.g., serum creatinine > 1.8 mg/dl)
9. Concomitant Urinary Tract Infection (UTI)
10. Concomitant bladder stones
11. Confirmed or suspected prostate/bladder cancer
12. Previous pelvic irradiation or radical pelvic surgery
13. Previous prostate surgery, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate
14. Chronic prostatitis, or recurring prostatitis within the past 12 months
15. Serious concurrent medical conditions such as uncontrolled diabetes
16. Known allergy to nickel
17. Life expectancy less than 12 months
18. Use of concomitant medications (e.g., anticholinergics, antispasmodics or antidepressants) affecting bladder function
19. Anti-coagulant, anti-platelet, or thrombolytic medication other than Acetylsalicylic Acid (ASA) or Clopidogrel. ASA and Clopidogrel must be ceased 7 days prior to the procedure.
20. 5--reductase inhibitors within 6 months of pre-treatment evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study).
21. -blockers within 2 weeks of pre-treatment evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued for entrance into or throughout the study).
22. Future fertility concerns
23. Any severe illness that might prevent study completion or would confound study results

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Device Success defined as both 1) deliverability of the implant and 2) freedom from unanticipated adverse events (UAEs) not listed in the protocol or AEs that meet the protocol definition of Serious AEs. | Intraoperative
  Frequency of Device Success is assessed by subject, for both successful device placement in the target anatomy and absence of serious or unanticipated adverse events through discharge.
Occurrence of device and/or procedure related Adverse Events as determined by investigator and independent medical reviewer | Intraoperative
  Frequency and severity of any device or procedure related adverse events, by subject.
Occurrence of Adverse Event specific to indwelling catheterization, descriptive analysis | Seven days following implantation of the investigational device
  Frequency of indwelling catheterization = or > 7 days following placement of the investigational device.
Effectiveness of implant measured through symptom improvement (International Prostate Symptom Score - IPSS) | 3 months following device placement
  Subjects should demonstrate improvement of > or = to 3 point reduction from baseline measurement.

SECONDARY OUTCOMES:
Assessment of Sexual Health using the Sexual Health in Men (SHIM) questionnaire | 6 months, 12-,24-,36-, months post implantation
  Observational assessment of subject scores on SHIM at the 6 months and 12 months visit, compared to baseline.
Assessment of Incontinence, using the Incontinence Severity Index (ISI) questionnaire | 2 weeks, 1 month, 3 months
  Observational assessment of subject scores on ISI at 2 weeks, 1 month and 3 months compared to baseline.
Observation of pain using a validated Visual Analogue Scale (VAS) questionnaire | through 3 month follow-up
  Observational assessment of subject reports of pain on the VAS questionnaire, at discharge and follow up visits up to 3 months, compared to baseline.
Improvement in Uroflowmetry compared to baseline | 3-, 6-, 12-, 24-, 36-months post implantation
  Uroflowmetry is measured at 3 months post implantation and compared to baseline
Effectiveness of implant measured through symptom improvement (International Prostate Symptom Score - IPSS) | 12 months 24 months and 36 months
  Observation of IPSS scores compared to baseline at 12 months follow up.
Effectiveness of the treatment by assessing need for further treatment to alleviate symptoms of BPH. | 12 months 24 months and 36 months
  Observation of incidence of repeat invasive treatment for LUTS through 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gilling, MD, Principal Investigator — Tauranga Urology Research Ltd.
Locations (3):
- MBAL "Tokuda Bolnitsa Sofia" AD, Sofia, Bulgaria
- New Zealand (2):
  - RoundHay Medical Center, Nelson South, Nelson Region
  - Tauranga Urology Research Ltd, Tauranga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Charles J, Valenti L, Britt H. BPH - management in general practice. Aust Fam Physician. 2011 Oct;40(10):757. PMID 22003475
- [Background] Woo HH, Gillman MP, Gardiner R, Marshall V, Lynch WJ. A practical approach to the management of lower urinary tract symptoms among men. Med J Aust. 2011 Jul 4;195(1):34-9. doi: 10.5694/j.1326-5377.2011.tb03185.x. PMID 21728939
- [Background] Milani S, Djavan B. Lower urinary tract symptoms suggestive of benign prostatic hyperplasia: latest update on alpha-adrenoceptor antagonists. BJU Int. 2005 Jun;95 Suppl 4:29-36. doi: 10.1111/j.1464-410X.2005.05485.x. PMID 15871733
- [Background] Schelin S, Geertsen U, Walter S, Spangberg A, Duelund-Jacobsen J, Kroyer K, Hjertberg H, Vatne V, Richthoff J, Nordling J. Feedback microwave thermotherapy versus TURP/prostate enucleation surgery in patients with benign prostatic hyperplasia and persistent urinary retention: a prospective, randomized, controlled, multicenter study. Urology. 2006 Oct;68(4):795-9. doi: 10.1016/j.urology.2006.05.020. PMID 17070355
- [Background] Bruskewitz RC, Larsen EH, Madsen PO, Dorflinger T. 3-year followup of urinary symptoms after transurethral resection of the prostate. J Urol. 1986 Sep;136(3):613-5. doi: 10.1016/s0022-5347(17)44991-3. PMID 2426477
- [Background] Thomas JA, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Bachmann A. A Multicenter Randomized Noninferiority Trial Comparing GreenLight-XPS Laser Vaporization of the Prostate and Transurethral Resection of the Prostate for the Treatment of Benign Prostatic Obstruction: Two-yr Outcomes of the GOLIATH Study. Eur Urol. 2016 Jan;69(1):94-102. doi: 10.1016/j.eururo.2015.07.054. Epub 2015 Aug 15. PMID 26283011
- [Background] Reich O, Gratzke C, Bachmann A, Seitz M, Schlenker B, Hermanek P, Lack N, Stief CG; Urology Section of the Bavarian Working Group for Quality Assurance. Morbidity, mortality and early outcome of transurethral resection of the prostate: a prospective multicenter evaluation of 10,654 patients. J Urol. 2008 Jul;180(1):246-9. doi: 10.1016/j.juro.2008.03.058. Epub 2008 May 21. PMID 18499179
- [Background] Mandeville J, Gnessin E, Lingeman JE. New advances in benign prostatic hyperplasia: laser therapy. Curr Urol Rep. 2011 Feb;12(1):56-61. doi: 10.1007/s11934-010-0153-1. PMID 21088938
- [Background] Ahyai SA, Lehrich K, Kuntz RM. Holmium laser enucleation versus transurethral resection of the prostate: 3-year follow-up results of a randomized clinical trial. Eur Urol. 2007 Nov;52(5):1456-63. doi: 10.1016/j.eururo.2007.04.053. Epub 2007 Apr 25. PMID 17499427
- [Background] Bachmann A, Tubaro A, Barber N, d'Ancona F, Muir G, Witzsch U, Grimm MO, Benejam J, Stolzenburg JU, Riddick A, Pahernik S, Roelink H, Ameye F, Saussine C, Bruyere F, Loidl W, Larner T, Gogoi NK, Hindley R, Muschter R, Thorpe A, Shrotri N, Graham S, Hamann M, Miller K, Schostak M, Capitan C, Knispel H, Thomas JA. 180-W XPS GreenLight laser vaporisation versus transurethral resection of the prostate for the treatment of benign prostatic obstruction: 6-month safety and efficacy results of a European Multicentre Randomised Trial--the GOLIATH study. Eur Urol. 2014 May;65(5):931-42. doi: 10.1016/j.eururo.2013.10.040. Epub 2013 Nov 11. PMID 24331152
- [Background] Gao YA, Huang Y, Zhang R, Yang YD, Zhang Q, Hou M, Wang Y. Benign prostatic hyperplasia: prostatic arterial embolization versus transurethral resection of the prostate--a prospective, randomized, and controlled clinical trial. Radiology. 2014 Mar;270(3):920-8. doi: 10.1148/radiol.13122803. Epub 2013 Nov 13. PMID 24475799
- [Background] Bouza C, Lopez T, Magro A, Navalpotro L, Amate JM. Systematic review and meta-analysis of Transurethral Needle Ablation in symptomatic Benign Prostatic Hyperplasia. BMC Urol. 2006 Jun 21;6:14. doi: 10.1186/1471-2490-6-14. PMID 16790044
- [Background] Roehrborn CG, Rukstalis DB, Barkin J, Gange SN, Shore ND, Giddens JL, Bolton DM, Cowan BE, Cantwell AL, McVary KT, Te AE, Gholami SS, Moseley WG, Chin PT, Dowling WT, Freedman SJ, Incze PF, Coffield KS, Borges FD, Rashid P. Three year results of the prostatic urethral L.I.F.T. study. Can J Urol. 2015 Jun;22(3):7772-82. PMID 26068624
- [Background] Peyton CC, Badlani GH. The management of prostatic obstruction with urethral stents. Can J Urol. 2015 Oct;22 Suppl 1:75-81. PMID 26497347
- [Background] Oesterling JE. A permanent, epithelializing stent for the treatment of benign prostatic hyperplasia. Preliminary results. J Androl. 1991 Nov-Dec;12(6):423-8. PMID 1722799
- [Background] Perry MJ, Roodhouse AJ, Gidlow AB, Spicer TG, Ellis BW. Thermo-expandable intraprostatic stents in bladder outlet obstruction: an 8-year study. BJU Int. 2002 Aug;90(3):216-23. doi: 10.1046/j.1464-410x.2002.02888.x. PMID 12133055
- [Background] Shore ND, Dineen MK, Saslawsky MJ, Lumerman JH, Corica AP. A temporary intraurethral prostatic stent relieves prostatic obstruction following transurethral microwave thermotherapy. J Urol. 2007 Mar;177(3):1040-6. doi: 10.1016/j.juro.2006.10.059. PMID 17296408
- [Background] Yildiz G, Bahouth Z, Halachmi S, Meyer G, Nativ O, Moskovitz B. Allium TPS--A New Prostatic Stent for the Treatment of Patients with Benign Prostatic Obstruction: The First Report. J Endourol. 2016 Mar;30(3):319-22. doi: 10.1089/end.2015.0593. Epub 2015 Nov 17. PMID 26472166
- [Background] Song HY, Kim CS, Jeong IG, Yoo D, Kim JH, Nam DH, Bae JI, Park JH. Placement of retrievable self-expandable metallic stents with barbs into patients with obstructive prostate cancer. Eur Radiol. 2013 Mar;23(3):780-5. doi: 10.1007/s00330-012-2650-8. Epub 2012 Sep 16. PMID 22983316
- [Background] Armitage JN, Cathcart PJ, Rashidian A, De Nigris E, Emberton M, van der Meulen JH. Epithelializing stent for benign prostatic hyperplasia: a systematic review of the literature. J Urol. 2007 May;177(5):1619-24. doi: 10.1016/j.juro.2007.01.005. PMID 17437773